CLINICAL TRIAL: NCT01734317
Title: An Open, Non Controled, Single-centre, Clinical Investigation to Evaluate Efficacy in Second Degree (Superficial, Deep or Mixed) Partial Thickness Burns When Using a Soft Silicone Wound Contact Ayer Containing Silver.
Brief Title: An Open Single-centre Investigation Evaluating Efficacy in Second Degree Partial Thickness Burns Using a Silicone Contact Layer Containing Silver.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MxT Ag 02
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2013-02

CONDITIONS: Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dressing (Experimental): Mepilex Transfer Ag is a soft silicone wound contact layer that absorbs and transfers exudate, maintains a moist wound healing environment and has antimicrobial properties.
  Interventions: Device: Mepilex Transfer Ag

INTERVENTIONS:
Device: Mepilex Transfer Ag — A soft silicone wound contact layer.

SUMMARY:
Approximately 10 subjects from one clinic having sustained a burn injury covering 1-25% or the Total Body surface Area (TBSA)and assessed as superficial partial-thickness or superficial deep-partial-thickness. The subject will be assessed once a week for a maximum of 3 weeks or until the burn is healed if that occurs earlier. . The dressing Mepilex Transfer Ag will be used as wound contact layer and gauze rolls and compression as second dressing.

DETAILED DESCRIPTION:
Approximately 10 subjects from one site will be evaluated provided they fulfill the inclusion criteria and none of the exclusion criteria and gives a signed and dated consent.

Subjects may have sustained a burn injury covering 1-25% of the Total Body Surface Area (TBSA)and assessed as superficial partial-thickness or superficial deep-partial thickness in dept. Each subject will be followed one time per week for a maximum of 3 weeks or until the burn is healed if that occurs earlier. Healing is defined as ≥95% epithelialisation. Percent (%) healed epithelialization will be measured by photo analysing using the PictZar program. Dressing changes will be performed at each visit and in between if deemed necessary by the investigator.Gauze rolls and compression will be used as secondary dressing.All dressing changes will be registered in a log. Pain before, during and after removal will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a second degree (superficial, deep or mixed) partial thickness burn from 1-25% TBSA.
* One single, isolated burn area selected for study site Study site area should be between 1-15% BSA
* Male or female
* From 18 years and above
* Either in- or out-patient
* Thermal burn injury
* Signed Informed Consent/Assent Form

Exclusion Criteria:

* Electrical, chemical burn etiology
* If any full thickness areas are present, these should not be > 5 %
* Burn greater than 36 hrs old
* Burns to face
* Use of chemical/enzymatic and biological debridement within 7 days of investigation start
* Presence of inflammation or infection in burn wounds
* Use of topical antibiotics, antiseptics, or antimicrobials in conjunction with study product.
* Subjects with lung injury or Subject being on a ventilator
* Subjects with dermatologic skin disorders or necrotizing processes
* Subjects with insulin dependent diabetes mellitus judged by the investigator to be a potential interference in the treatment
* Diagnosed underlying disease(s) (e.g HIV/AIDS, cancer and severe anaemia) judged by the investigator to be a potential interference in the treatment
* Subject not expected to follow the investigation procedures
* Subjects previously included in this investigation
* Subjects included in other ongoing clinical investigation at present or during the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Schweiger, MD, Principal Investigator — Florida Gulf-toBay Anesthesiology, Tampa Bay Circle
Locations (2):
- United States (2):
  - Florida Gulf-to-bay Anesthesiology, Tampa, Florida
  - Long Island Plastic Surgical Group, P.C, Garden City, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dressing
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mepilex Transfer Ag
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Healing
Description: Healing at day 14 pt 21. Healing was defined as ≥95% epithelialisation. The PictZar program will be used to analyze burn wound healing by tissue type. ("The PictZar equipment for this analysis will be located at MHC HQ, however, the analysis will be performed by a clinician not affiliated with MHC.") Each subject was followed/assessed one time per week for a maximum of 3 weeks or until the burn was healed if that occured earlier.
Time Frame: 14 days and 21 days
Measure: Number; unit: participants
Arm/Group | Dressing
Number analyzed (Participants) | 10
participants | 10

2. Secondary Outcome: Baseline (Visit 1) Pain Will be Measured Before Burn Assessment Visit 2-3, Pain Will be Measured (Pain BEFORE Dressing Removal, DURING Dressing Removal, AFTER Dressing Removal, 30 Min After Removal
Description: Pain will be measured by using the VAS scale, by placing a vertical mark across the 100 mm long horizontal line, from No pain to the left to Most intense pain imaginable to the right.
  Baseline (Visit 1) Pain will be measured before burn assessment Visit 2-4, Pain will be measured (Pain BEFORE dressing removal, DURING dressing removal, AFTER dressing removal, 30 min after removal
Time Frame: After 0/14/21 days treatment
Population: No data collected
Arm/Group | Pain Measure
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Dressing
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other